CLINICAL TRIAL: NCT03742869
Title: A Multi-omics Study on the Human Papillomavirus Integration and Tumorigenesis of Uterine Cervical Adenocarcinoma
Brief Title: HPV Integration and Tumorigenesis of Uterine Cervical Adenocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: HITA
Record Dates: First submitted 2018-11-09; First posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Cervical Adenocarcinoma; Human Papillomavirus; Genome-wide Association Study; Whole Exome Sequencing; Transcriptome; Metabolome; Tumorigenesis; Prognosis
MeSH Terms: conditions — Carcinogenesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — An 8 ml peripheral venous blood, and 50 μL cancer tissue and tissue adjacent to cancer will be collected from eligible patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with HPV integration: The HPV integration status will be checked by GWAS.
  Interventions: Combination Product: A multi-omics analysis
- Patients without HPV integration: The HPV integration status will be checked by GWAS.
  Interventions: Combination Product: A multi-omics analysis

INTERVENTIONS:
Combination Product: A multi-omics analysis — A multi-omics analysis including genome-wide association study, whole exome sequencing, transcriptomics and metabolomics.

SUMMARY:
This study aims to analyze the multi-omics results between uterine cervical adenocarcinoma patients with and without human papillomavirus (HPV) infections. The multi-omics profiles include genome wide association study (GWAS), whole exome sequencing, analysis of transcriptomics and metabolomics. The HPV integration status is interpreted by GWAS. A comprehensive multi-omics will reveal the role of HPV integration in the molecular mechanism of tumorigenesis and prognosis of uterine cervical adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed primary adenocarcinoma of the uterine cervix
* Signed an approved informed consents
* Feasible for biopsy

Exclusion Criteria:

* Not meeting all of the inclusion criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients confirmed primary adenocarcinoma of the uterine cervix
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-11-10 (Actual); Primary Completion 2021-11-23 (Estimated); Study Completion 2021-11-23 (Estimated)

PRIMARY OUTCOMES:
Frequencies of somatic driving mutations | Two years
  The differences of frequencies of somatic driving mutations will be compared between patients with and without HPV integration.

SECONDARY OUTCOMES:
Frequencies of alteration of RNA expression | Two years
  The alteration of patterns of RNA expression, including mRNA, miRNA, and lncRNA, will be compared between patients with and without HPV integration.
Frequencies of alteration of protein expression and signal pathway | Two years
  The alteration of patterns of protein expression and signal pathway will be compared between patients with and without HPV integration.
Progression-free survival | Five years
  Progression-free survival between patients with differential expressed multi-omics will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All data will be available to all researchers.
Supporting Information: CSR
Time Frame: All data will be available to all researchers once related papers have been accepted publicly, and will be available for ever.